CLINICAL TRIAL: NCT00241540
Title: Efficacy of Esomeprazole 40 mg Once Daily Versus Placebo & Esomeprazole 20 mg Once Daily Versus Placebo in Treatment for Relief of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs Including COX-2 Selective NSAIDs
Brief Title: Esomeprazole for Relief of Upper Gastrointestinal Symptoms Associated With Continuous Use of NSAIDs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9617C00001; SH-NEN-0001
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: GERD
Keywords: NSAIDs; Upper GI symptoms
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
This study is a randomised, double-blind, parallel-group and placebo controlled study comparing the efficacy of esomeprazole 40 mg orally qd vs. placebo and esomeprazole 20 mg orally qd vs. placebo when given to patients on continuous use of NSAIDs, including COX-2 selective NSAIDs, for a period of 4 weeks in treatment of relief of upper GI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, or older.
* Capable of completing the diary card.
* Ability to complete the HRQL questionnaires.
* A clinical diagnosis of a chronic condition (e.g., osteoarthritis or rheumatoid arthritis) that requires continuous daily NSAID treatment for at least 7 months.
* Daily NSAID treatment is defined as taking the prescribed dose for at least 5 of 7 days in any given week and can include COX-2 selective NSAIDs, multiple NSAIDs, and high-dose aspirin (>325 mg/day).
* Daily NSAID treatment dose and type: (Must have been stable for at least 4 weeks prior to baseline endoscopy and; Are expected to remain stable for the duration of the study. and; Must be administered orally for the duration of the study. If more than one type of NSAID treatment is used, at least one type must be given orally).

Exclusion Criteria:

* Current, or history of, gastric or duodenal ulcer
* Current, or history of, esophageal, gastric or duodenal surgery.
* History of GERD, not associated with NSAID use.
* Pain, discomfort or burning in the upper abdomen precipitated by exercise or relieved by defecation.
* Pain, discomfort or burning in the upper abdomen not associated with the use of NSAIDs, including COX-2 selective NSAIDs, as judged by the investigator.
* Endoscopic Barrett's esophagus(>3 cm) or significant dysplastic changes in the esophagus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808
Dates: Start 2001-01; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of esomeprazole versus placebo through 4 weeks of treatment of upper GI symptoms associated with nonsteroidal anti-inflammation

SECONDARY OUTCOMES:
- To assess the safety & tolerability of esomeprazole versus placebo when administered for up to 4 weeks to patients receiving daily NSAID therapy
- To assess the impact of treatment

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Nexium Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (119):
- United States (19):
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, South Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Conyers, Georgia
  - Research Site, Newburgh, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Tulsa, Oklahoma
  - Research Site, Tipton, Pennsylvania
  - Research Site, Norfolk, Virginia
  - Research Site, Virginia Beach, Virginia
- Belgium (35):
  - Research Site, Alleur
  - Research Site, Ans
  - Research Site, Beernem
  - Research Site, Betekom
  - Research Site, Bottelare
  - Research Site, Braine-l'Alleud
  - Research Site, Brussels (Ixelles)
  - Research Site, Brussels (Jette)
  - Research Site, Brussels (Uccle)
  - Research Site, Buizingen
  - Research Site, Duffel
  - Research Site, Durnal
  - Research Site, Erembodegem
  - Research Site, Forest
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Halle
  - Research Site, Herentals
  - Research Site, Lambermont
  - Research Site, Leut
  - Research Site, Liège
  - Research Site, Linkebeek
  - Research Site, Maasmechelen
  - Research Site, Massemen
  - Research Site, Merelbeke
  - Research Site, Natoye
  - Research Site, Nivelles
  - Research Site, Oud-Heverlee
  - Research Site, Seraing
  - Research Site, Soignies
  - Research Site, Uccle
  - Research Site, Vorst (Brussels)
  - Research Site, Waremme
  - Research Site, Zoersel
  - Research Site, Zolder
- France (19):
  - Research Site, Albens
  - Research Site, Angers
  - Research Site, Dambach-la-Ville
  - Research Site, Dommartin-les-touls
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Gesté
  - Research Site, Gémenos
  - Research Site, Husseren-Wesserling
  - Research Site, La Regrip
  - Research Site, Le Pian-Médoc
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Maromme
  - Research Site, Mont-de-Marsan
  - Research Site, Montingy Les Metz
  - Research Site, Paris
  - Research Site, Saint-Ouen
  - Research Site, Strasbourg
  - Research Site, Tarare
- Germany (27):
  - Research Site, Berlin
  - Research Site, Bernau
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Genthin
  - Research Site, Herne
  - Research Site, Kelkheim
  - Research Site, Künzing
  - Research Site, Lienen
  - Research Site, Lüdenscheid
  - Research Site, München
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Passau
  - Research Site, Potsdam
  - Research Site, Ratingen
  - Research Site, Regensburg
  - Research Site, Ribnitz-Damgarten
  - Research Site, Saarbrücken
  - Research Site, Salzgitter
  - Research Site, Stockach
  - Research Site, Wangen
  - Research Site, Wiesbaden
  - Research Site, Wolmirstedt
- Hungary (7):
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Dunaújváros
  - Research Site, Szentes
  - Research Site, Szombathely
  - Research Site, Vác
  - Research Site, Veszprém
- Spain (12):
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, Guadalajara
  - Research Site, Madrid
  - Research Site, Mérida
  - Research Site, Palma de Mallorca
  - Research Site, San Sebastián(Guipuzcoa)
  - Research Site, Seville
  - Research Site, Torrelavega
  - Research Site, Valencia
  - Research Site, Viladecans
  - Research Site, Zaragoza